CLINICAL TRIAL: NCT05428618
Title: The Effect of Mobile Support Application Developed for Patients Undergoing Bariatric Surgery on Self-Management, Quality of Life and Clinical Outcomes
Brief Title: Mobile Application for Bariatric Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Damla Seckin, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: w34dsxfh
Record Dates: First submitted 2022-02-10; First posted 2022-06-23 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2023-09

CONDITIONS: Obesity; Bariatric Surgery; Quality of Life; Complication; Mobile Health; EHealth; Self Management
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- e-BariS app Group (Experimental): "Self-Monitoring Module" and "Patient Education Module"
  Interventions: Other: e-BariS app group
- Self-Monitoring Group (Sham Comparator): "Self-Monitoring Module"
  Interventions: Other: Self-Monitoring Group

INTERVENTIONS:
Other: e-BariS app group — During the discharge process, informed consent will be obtained from the patients and the measurement tools will be filled and the mobile application will be downloaded to their phones. The intervention group will have access to all the content of the mobile application, which includes the "Self-Monitoring Module" and the "Patient Education Module". Passwords will be defined so that patients in the intervention group can access the "Patient Education Module". Information on the introduction and use of the application will be presented to the patient by the researcher.
  The patients will be followed for six months within the scope of the project. In addition, reminder notifications will be sent to patients via the mobile application in line with the areas that patients can access. At one, three, and six months after surgery, he will complete other assessment scales during outpatient follow-up. For patients providing remote control, the scale will be sent online.
  Arms: e-BariS app Group
Other: Self-Monitoring Group — Patients in the control group will only have access to the "Self-Monitoring Module" in the application. Other fields will be encrypted. Patients in the control group will also be informed about the area they can access. Patients in the control group will only have access to the self-monitoring section. One, three, and six months after surgery, she will complete other assessment scales during her outpatient follow-up. Scales will be sent online for patients providing remote control. After the project is completed, all content will be opened to the control group patients.
  Arms: Self-Monitoring Group

SUMMARY:
Introduction: One of the alternative ways, as a result of the increasing demand for health services and the inadequacy of meeting the increasing needs, is mobile health applications. According to TUIK 2019 data, the rate of having mobile phones in households is 98.7%. With the development of technology, all information can be integrated into the mobile phone, and mobile applications allow the patient to give data from the environment in which he lives and to evaluate himself. Self-assessment and monitoring of the patient enable the patient to participate in his/her self-care, supports self-management behaviors, and improves their quality of life.

Objective: It was aimed to develop a mobile support application for patients undergoing bariatric surgery and to evaluate the effect of application use on patients' self-management, quality of life, and clinical outcomes.

Method: In the first stage;

* Preparing the information to be included in the mobile health application that is planned to be developed and evaluating the quality of the content,
* Parallel to this, the adaptation of the "Bariatric Surgery Self-Management Behaviors Scale" into Turkish and the evaluation of its validity and reliability.
* Design of the mobile application, transferring the educational content to the mobile application,
* It is aimed to evaluate the technical suitability and usability of the mobile application.

In the second stage, it was aimed to conduct a randomized controlled study to determine the effect of the developed mobile application on the self-management, quality of life and clinical outcomes of the patients.

The developed mobile application will be introduced to patients at discharge after bariatric surgery. Rating scales will be administered to patients at the end of one, three, and six months after surgery. These scales are the Bariatric Surgery Self-Management Behaviors Scale and the Moorehead-Ardelt Quality of Life Scale-II.

Conclusion: It is expected that the mobile application-based education to be developed for bariatric surgery will improve the patients' post-surgical self-management, increase their quality of life and decrease the early complication rates.

ELIGIBILITY:
Inclusion Criteria:

* Speaking and understanding Turkish,
* Being literate
* Having the ability to use a smartphone,
* Having a mobile phone with IOS or Android software,
* Having internet access,
* Having consented to download the mobile application to the mobile phone,
* Between the ages of 18-65,
* Patients undergoing bariatric surgery for the first time.

Exclusion Criteria:

* Patients with vision or hearing problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Self-Management | Change from baseline BBSQ at one month, Change from baseline BBSQ at 3 months, Change from baseline BBSQ at 6 months
  The self-management scores of the patients will be measured with the Bariatric Surgery Self-Management Behaviors Scale.
  The scale was developed by Welch and colleagues in 2008. Validity and reliability were done in Iran in 2018.
  It consists of seven factors and 33 items, including eating behaviors (8), fluid intake (8), physical activity (3), dumping syndrome management (4), vitamin and mineral supplement (4), fruit, vegetable, and cereals (3), protein intake (3). It is evaluated with a triple Likert scale as never, sometimes, and always. Subscale and total scores were converted to the range of 0-100, higher scores indicate higher self-management.
Quality of Life Scale | Change from baseline MA-II at one month, Change from baseline MA-II at 3 months, Change from baseline MA-II at 6 months
  The Moorehead-Ardelt Quality of Life Scale (MA-II) was developed in 1998. The scale consists of six questions including self-esteem, physical function, social relations, ability to work, sexuality, and eating behavior. At the same time, each item of the scale is supported by figures related to the subject in order to help individuals from different cultures understand. Each item has a 10-point Likert-type measure. Each item is equally weighted and increases and decreases by 0.10 points positively and negatively, keeping the 0 value in the center. While each item decreases by 0.10 points from the "0" point to the left, it increases by 0.10 points to the right. The scores for each item range from -0.50 to 0.50. The total scale scoring varies between -3 and +3, the score between -2.1 and -3 is considered a very poor quality of life, and between +2.1 and +3, the quality of life is considered.

SECONDARY OUTCOMES:
Weight loss | Change from baseline kilogram for weight loss at one month, Change from baseline kilogram for weight loss at 3 months, Change from baseline kilogram for weight loss at 6 months
  Official measurements made by the hospital Measurements will be made in kg
Nausea | Change from baseline Visual Analog Scale (VAS) for nausea at one month, Change from one month VAS for nausea at 3 months, Change from 3 months VAS for nausea at 6 months
  Nausea after eating will be questioned in the evaluation of dumping syndrome. Nausea will be evaluated with a self-reported scale the Visual Analog Scale. The scale ranges from 1 to 10. In the measurement, 1 = I have no nausea, 10 = I have unbearable nausea.
Vomiting | Change from baseline Visual Analog Scale (VAS) for vomiting at one month, Change from one month VAS for vomiting at 3 months, Change from 3 months VAS for vomiting at 6 months
  Vomiting after eating will be questioned in the evaluation of dumping syndrome. Vomiting will be evaluated with a self-reported scale the Visual Analog Scale. The scale ranges from 1 to 10. In the measurement, 1 = I have no vomiting, 10 = I have unbearable vomiting.
Dizziness | Change from baseline Visual Analog Scale (VAS) for dizziness at one month, Change from one month VAS for dizziness at 3 months, Change from 3 months VAS for dizziness at 6 months
  Dizziness after eating will be questioned in the evaluation of dumping syndrome.
  Dizziness will be evaluated with a self-reported scale the Visual Analog Scale. The scale ranges from 1 to 10. In the measurement, 1 = I have no dizziness, 10 = I have unbearable dizziness.
Pain-Visual Analog Scale | Change from baseline Visual Analog Scale (VAS) for pain at one month, Change from one month VAS for pain at 3 months, Change from 3 months VAS for pain at 6 months
  Pain will be evaluated with a self-reported scale the Visual Analog Scale. The scale ranges from 1 to 10. In the measurement, 1 = I have no pain, 10 = I have unbearable pain.
wound infection | Change from baseline Visual Analog Scale (VAS) for wound infection at one month.
  Wound infection will be evaluated with a self-reported scale the Visual Analog Scale. The scale ranges from 1 to 10. In the measurement, 1 = I have no wound infection, 10 = I have an unbearable wound infection.
Hypoglycemia | Change from baseline Visual Analog Scale (VAS) for hypoglycemia at one month, Change from one month VAS for hypoglycemia at 3 months, Change from 3 months VAS for hypoglycemia at 6 months.
  Hypoglycemia will be evaluated with a self-reported scale the Visual Analog Scale. The scale ranges from 1 to 10. In the measurement, 1 = I have no hypoglycemia, 10 = I have unbearable hypoglycemia.
Constipation | Change from baseline Visual Analog Scale (VAS)for constipation at one month, Change from one month VAS for constipation at 3 months, Change from 3 months VAS for constipation at 6 months.
  Constipation will be evaluated with a self-reported scale the Visual Analog Scale. The scale ranges from 1 to 10. In the measurement, 1 = I have no constipation, 10 = I have unbearable constipation.
Number of emergency admissions | Change from baseline Number of emergency admissions at one month, Change from one month number of emergency admissions at 3 months, Change from 3 months number of emergency admissions at 6 months.
  A number of emergency admissions will be evaluated with a self-reported. How many times the patient applied to the emergency department will be evaluated by asking open-ended questions.
Number of hospital readmission | Change from baseline number of hospital readmission at one month, Change from one month number of hospital readmission at 3 months, Change from 3 months number of hospital readmission at 6 months.
  A number of hospital readmission will be evaluated with a self-reported. How many times the patient applied to the emergency department will be evaluated by asking open-ended questions.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Antalya, Antalya
  - Hospital, Antalya

IPD SHARING:
Plan to Share IPD: No